CLINICAL TRIAL: NCT04048577
Title: The Impact of a Planned 12-week Dosing Interruption of Natalizumab on Immune Cell Trafficking, Pharmacokinetic (PK)/Pharmacodynamic (PD) Parameters, and Multiple Sclerosis (MS) Disease Stability.
Brief Title: A Pilot Study to Characterize the Biological Effect of a Pre-planned 12 Week Dose Interruption of Natalizumab
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Berkovich, Regina MD, PhD Inc. (Other)
Collaborators: Biogen (Industry); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Regina Radner Berkovich, Director, Berkovich, Regina MD, PhD Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001-BIO-CSF
Record Dates: First submitted 2019-04-15; First posted 2019-08-07 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting
Keywords: Natalizumab; Drug Holiday; Alternative Dosing; Extended Dosing
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Interruption (Experimental): All subjects will continue to receive their prescribed Tysabri® 300 mg IV infusions at their approved infusion sites. The patients will receive Tysabri at standard intervals (28-days) except during the pre-planned dose interruption of 2 consecutive skipped doses.
  Interventions: Drug: Dosing Interruption of Natalizumab
- Standard Treatment (No Intervention): All subjects will continue to receive their prescribed Tysabri® 300 mg IV infusions at their approved infusion sites. The patients will receive Tysabri at standard intervals (28-days).

INTERVENTIONS:
Drug: Dosing Interruption of Natalizumab — Planned 12 week dosing interruption of natalizumab
  Other Names: Dosing Interruption of Tysabri
  Arms: Dose Interruption

SUMMARY:
This is an open-label study of patients with relapsing forms of MS is designed to assess the biochemical, immunological, and kinetic profiles of natalizumab being used with specific brief dosing interruption. The study will be conducted at one site in the US. Ten subjects currently treated with natalizumab will be enrolled and will be evaluated for both PK/PD and cell trafficking in blood and/or CSF during standard dosing of natalizumab and at the end of a planned 12-week dosing interruption. MS disease activity will be carefully monitored clinically and by MRI and NfL.

DETAILED DESCRIPTION:
Study Title:

The impact of a planned 12-week dosing interruption of natalizumab on immune cell trafficking, PK/PD parameters, and MS disease stability.

Objectives:

Hypothesis: An interruption in the dosing of natalizumab results in a lower risk of progressive multifocal leukoencephalopathy (PML) while maintaining MS disease control by selective immune surveillance.

Primary endpoints: To measure the re-establishment of immune surveillance by measuring leukocyte cell binding to the blood brain barrier and trafficking into the central nervous system (CNS) during a planned 12-week dosing interruption of natalizumab. This will be done by measuring leukocytes in the CSF. Concurrently, MS disease activity will be monitoring with MRI.

Secondary endpoints:

* To characterize the difference in PK/PD parameters in patients during standard 28-day dosing intervals vs. at the end of a planned 12-week dosing interruption
* To measure natalizumab drug concentrations, Soluble Vascular Cell Adhesion Molecule (sVCAM), Soluble Mucosal Vascular Addressin Cell Adhesion Molecule (sMAdCAM), Very Late Antigen-4 (VLA4) expression, and receptor occupancy measured in blood.
* To measure neurofilament light (NfL) in CSF and serum as a sensitive measure of MS disease stability.
* Using MRI and clinical parameters, to determine impact of a planned 12-week dosing interruption of natalizumab on MS disease stability.
* MRI's will be obtained for each patient at the end of the dose interruption and 3 months after the re-initiation of natalizumab dosing.

Design:

Single site, open-label, consenting patients with relapsing forms of Multiple Sclerosis who are scheduled for a dose interruption of natalizumab. Patients will provide biological samples (blood and CSF) and have MRIs post-dose interruption.

Patient Population:

Patients with relapsing forms of Multiple Sclerosis who are currently on natalizumab therapy with stable MS disease and who are scheduled for a planned 12-week dosing interruption.

Treatment Groups:

Duration of Study Participation: Up to 9 months Study Location: 8727 Beverly Blvd, West Hollywood, California (CA) 90048 United States (US) Study Phase: Pilot exploratory study. Number of Planned Subjects: 10 Sample Size Determination: This is an exploratory study. No formal sample size calculation was performed.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for entry into this study, candidates must meet all of the following eligibility criteria at the time of randomization:

Screening Visit:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
2. At least 18 years old at the time of informed consent.
3. Must be a patient with a relapsing form of Multiple Sclerosis enrolled in the TOUCH Prescribing Program who is not expected to discontinue Tysabri® therapy prior to completion of the requirements of this study.
4. Must weigh between 50 and 110 kg, inclusive.
5. Patients must be considered clinically stable and scheduled for their pre-planned annual dose interruption of 2 consecutive skipped doses.
6. No evidence of disease activity with on standard (28-day interval) dosing of natalizumab.

Exclusion Criteria:

Candidates will be excluded from study entry if any of the following exclusion criteria exist at the time of screening:

Medical History

1. If subject answers 'Yes" to any question on the PML questionnaire that is not resolved prior to infusion as per standard operating procedure for natalizumab infusion.
2. If subject consumes alcohol within 24 hours of blood specimen collection.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Leukocyte Type and Quantity in CSF | Change of Leukocyte types and quantity in CSF in pre- and post-interruption of treatment through study completion, an average of 6 months.
  Types and quantities of leukocytes including T-cells, B-cells, macrophages, monocytes, etc. measured through flow cytometry.
MS Activity through CSF, Blood, and MRI | Change of MS Activity in pre- and post-interruption of treatment through study completion, an average of 6 months.
  Soluble factors related to MS activity include Neurofilament Light Chain Levels in Blood and CSF measured through flow cytometry. MRI of brain, cervical, and thoracic cavity will be closely monitored for MS disease activity.

SECONDARY OUTCOMES:
Natalizumab Concentrations in Blood | Change of Natalizumab Concentrations in Blood in pre- and post-interruption of treatment through study completion, an average of 6 months.
immunoglobulin G4 Levels in Blood | Change of immunoglobulin G4 Levels in Blood in pre- and post-interruption of treatment through study completion, an average of 6 months.
Soluble Vascular Cell Adhesion Molecules and Soluble Mucosal Vascular Addressin Cell Adhesion Molecule Levels (sVCAM sMAdCAM) in Blood | Change of sVCAM sMAdCAM in blood in pre- and post-interruption of treatment through study completion, an average of 6 months.
  sVCAM sMAdCAM are ligands that are released into the bloodstream as marker of inflammation. The measurements will be done with Luminex technology using VCAM1 and MAdCAM1 specific antibodies to measure the levels in serum.
John Cunningham Virus Extracellular Vesicle Antibody Levels in CSF | Change of John Cunningham Virus Extracellular Vesicles in CSF in pre- and post-interruption of treatment through study completion, an average of 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Regina R Berkovich, MD, PhD, Principal Investigator — Regina Berkovich MD, PhD Inc.
Locations (1):
- Regina Berkovich MD, PhD Inc., West Hollywood, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berkovich R, Togasaki DM, Cen SY, Steinman L. CD4 cell response to interval therapy with natalizumab. Ann Clin Transl Neurol. 2015 May;2(5):570-4. doi: 10.1002/acn3.190. Epub 2015 Mar 6. PMID 26000328
- [Background] Bloomgren G, Richman S, Hotermans C, Subramanyam M, Goelz S, Natarajan A, Lee S, Plavina T, Scanlon JV, Sandrock A, Bozic C. Risk of natalizumab-associated progressive multifocal leukoencephalopathy. N Engl J Med. 2012 May 17;366(20):1870-80. doi: 10.1056/NEJMoa1107829. PMID 22591293
- [Background] Disanto G, Barro C, Benkert P, Naegelin Y, Schadelin S, Giardiello A, Zecca C, Blennow K, Zetterberg H, Leppert D, Kappos L, Gobbi C, Kuhle J; Swiss Multiple Sclerosis Cohort Study Group. Serum Neurofilament light: A biomarker of neuronal damage in multiple sclerosis. Ann Neurol. 2017 Jun;81(6):857-870. doi: 10.1002/ana.24954. PMID 28512753
- [Background] Foley J, Zhovtis Ryerson L, Chang I, Kister I, Cutter G, Metzger R, Goldberg JD, Li X, Riddle E, Kasliwal R, Ren Z, Hotermans C, Ho PR, Campbell N. Progressive multifocal leukoencephalopathy occurring with extended interval dosing of natalizumab: Analysis of cases in the TOUCH database. CMSC 2018; 5698.
- [Background] Foley J, Metzger R, Hoyt T, Christensen A. Optimizing the natalizumab dose interval to reduce PML risk - lessons from the pharmacokinetics of therapy discontinuation. AAN 2015; P4.032.
- [Background] Ho PR, Koendgen H, Campbell N, Haddock B, Richman S, Chang I. Risk of natalizumab-associated progressive multifocal leukoencephalopathy in patients with multiple sclerosis: a retrospective analysis of data from four clinical studies. Lancet Neurol. 2017 Nov;16(11):925-933. doi: 10.1016/S1474-4422(17)30282-X. Epub 2017 Sep 29. PMID 28969984
- [Background] Khatri BO, Man S, Giovannoni G, Koo AP, Lee JC, Tucky B, Lynn F, Jurgensen S, Woodworth J, Goelz S, Duda PW, Panzara MA, Ransohoff RM, Fox RJ. Effect of plasma exchange in accelerating natalizumab clearance and restoring leukocyte function. Neurology. 2009 Feb 3;72(5):402-9. doi: 10.1212/01.wnl.0000341766.59028.9d. PMID 19188571
- [Background] Kuhle J, Kropshofer H, Haering DA, Kundu U, Meinert R, Barro C, Dahlke F, Tomic D, Leppert D, Kappos L. Blood neurofilament light chain as a biomarker of MS disease activity and treatment response. Neurology. 2019 Mar 5;92(10):e1007-e1015. doi: 10.1212/WNL.0000000000007032. Epub 2019 Feb 8. PMID 30737333
- [Background] Novakova L, Zetterberg H, Sundstrom P, Axelsson M, Khademi M, Gunnarsson M, Malmestrom C, Svenningsson A, Olsson T, Piehl F, Blennow K, Lycke J. Monitoring disease activity in multiple sclerosis using serum neurofilament light protein. Neurology. 2017 Nov 28;89(22):2230-2237. doi: 10.1212/WNL.0000000000004683. Epub 2017 Oct 27. PMID 29079686
- [Background] Plavina T, Subramanyam M, Bloomgren G, Richman S, Pace A, Lee S, Schlain B, Campagnolo D, Belachew S, Ticho B. Anti-JC virus antibody levels in serum or plasma further define risk of natalizumab-associated progressive multifocal leukoencephalopathy. Ann Neurol. 2014 Dec;76(6):802-12. doi: 10.1002/ana.24286. Epub 2014 Oct 24. PMID 25273271
- [Background] Plavina T, Muralidharan KK, Kuesters G, Mikol D, Evans K, Subramanyam M, Nestorov I, Chen Y, Dong Q, Ho PR, Amarante D, Adams A, De Seze J, Fox R, Gold R, Jeffery D, Kappos L, Montalban X, Weinstock-Guttman B, Hartung HP, Cree BAC. Reversibility of the effects of natalizumab on peripheral immune cell dynamics in MS patients. Neurology. 2017 Oct 10;89(15):1584-1593. doi: 10.1212/WNL.0000000000004485. Epub 2017 Sep 15. PMID 28916537
- [Background] Zhovtis Ryerson L, Foley J, Chang I, Kister I, Cutter G, Metzger R, Goldberg JD, Li X, Riddle E, Yu B, Ren Z, Hotermans C, Ho PR, Campbell N. Natalizumab extended interval dosing is associated with a reduction in progressive multifocal leukoencephalopathy risk in the TOUCH registry. ACTRIMS 2018; LB250.
- [Background] Zhovtis Ryerson L, Frohman TC, Foley J, Kister I, Weinstock-Guttman B, Tornatore C, Pandey K, Donnelly S, Pawate S, Bomprezzi R, Smith D, Kolb C, Qureshi S, Okuda D, Kalina J, Rimler Z, Green R, Monson N, Hoyt T, Bradshaw M, Fallon J, Chamot E, Bucello M, Beh S, Cutter G, Major E, Herbert J, Frohman EM. Extended interval dosing of natalizumab in multiple sclerosis. J Neurol Neurosurg Psychiatry. 2016 Aug;87(8):885-9. doi: 10.1136/jnnp-2015-312940. Epub 2016 Feb 25. PMID 26917698